CLINICAL TRIAL: NCT04798209
Title: A Single-center, Double-blind, Randomized, Placebo-controlled Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single- and Multiple-ascending Doses of ACT-777991 in Healthy Subjects
Brief Title: A Study to Examine the Safety, Tolerability, and Pharmacokinetics of Single- and Multiple-ascending Doses of ACT-777991 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-089-101; 2020-004464-26 (EudraCT Number)
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, randomized, placebo-controlled Phase 1 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Part A (single ascending dose) Dose A1 (Experimental): Single dose A1 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A2 (Experimental): Single dose A2 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A3 (Experimental): Single dose A3 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A4 (Experimental): Single dose A4 of ACT-777991 under fasted and fed conditions, separated by at least 14 days.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A5 (Experimental): Single dose A5 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A6 (Experimental): Single dose A6 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A7 (Experimental): Single dose A7 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part A (single ascending dose arm) Dose A8 (Experimental): Single dose A8 of ACT-777991.
  Interventions: Drug: ACT-777991 (SAD); Drug: Placebo (SAD)
- Part B (multiple ascending dose) Dose B1 (Experimental): Multiple doses B1 of ACT-777991.
  Interventions: Drug: ACT-777991 (MAD); Drug: Placebo (MAD)
- Part B (multiple ascending dose) Dose B2 (Experimental): Multiple doses B2 of ACT-777991.
  Interventions: Drug: ACT-777991 (MAD); Drug: Placebo (MAD)
- Part B (multiple ascending dose) Dose B3 (Experimental): Multiple doses B3 of ACT-777991.
  Interventions: Drug: ACT-777991 (MAD); Drug: Placebo (MAD)
- Part B (multiple ascending dose) Dose B4 (Experimental): Multiple doses B4 of ACT-777991.
  Interventions: Drug: ACT-777991 (MAD); Drug: Placebo (MAD)
- Part B (multiple ascending dose) Dose B5 (Experimental): Multiple doses B5 of ACT-777991.
  Interventions: Drug: ACT-777991 (MAD); Drug: Placebo (MAD)
- Part A (single ascending dose) Absolute Bioavailability (Experimental): Single dose of ACT-777991 plus a single dose of 14C-ACT-777991. At one of the dose levels from A4 to A8.
  Interventions: Drug: 14C-ACT-777991 microtracer (SAD - Absolute Bioavailability); Drug: Microtracer matching placebo (SAD - Absolute Bioavailability)
- Part B (multiple ascending dose) ADME (Experimental): Multiple doses of ACT-777991 plus a single dose of 14C-ACT-777991. At one of the dose levels from B1 to B5.
  Interventions: Drug: 14C-ACT-777991 microtracer (MAD - ADME); Drug: Microtracer matching placebo (MAD - ADME)

INTERVENTIONS:
Drug: ACT-777991 (SAD) — ACT-777991 administered as hard capsules for oral use.
  Arms: Part A (single ascending dose arm) Dose A2; Part A (single ascending dose arm) Dose A3; Part A (single ascending dose arm) Dose A4; Part A (single ascending dose arm) Dose A5; Part A (single ascending dose arm) Dose A6; Part A (single ascending dose arm) Dose A7; Part A (single ascending dose arm) Dose A8; Part A (single ascending dose) Dose A1
Drug: ACT-777991 (MAD) — ACT-777991 administered as hard capsules for oral use, once daily.
  Arms: Part B (multiple ascending dose) Dose B1; Part B (multiple ascending dose) Dose B2; Part B (multiple ascending dose) Dose B3; Part B (multiple ascending dose) Dose B4; Part B (multiple ascending dose) Dose B5
Drug: Placebo (SAD) — ACT-777991 matching placebo administered as hard capsules for oral use.
  Arms: Part A (single ascending dose arm) Dose A2; Part A (single ascending dose arm) Dose A3; Part A (single ascending dose arm) Dose A4; Part A (single ascending dose arm) Dose A5; Part A (single ascending dose arm) Dose A6; Part A (single ascending dose arm) Dose A7; Part A (single ascending dose arm) Dose A8; Part A (single ascending dose) Dose A1
Drug: Placebo (MAD) — Matching placebo administered as hard capsules for oral use, once daily.
  Arms: Part B (multiple ascending dose) Dose B1; Part B (multiple ascending dose) Dose B2; Part B (multiple ascending dose) Dose B3; Part B (multiple ascending dose) Dose B4; Part B (multiple ascending dose) Dose B5
Drug: 14C-ACT-777991 microtracer (SAD - Absolute Bioavailability) — Single dose of 14C-ACT-777991 microtracer, administered intravenously.
  Arms: Part A (single ascending dose) Absolute Bioavailability
Drug: Microtracer matching placebo (SAD - Absolute Bioavailability) — Single dose of 14C-ACT-777991 microtracer matching placebo, administered intravenously.
  Arms: Part A (single ascending dose) Absolute Bioavailability
Drug: 14C-ACT-777991 microtracer (MAD - ADME) — Single dose of 14C-ACT-777991 microtracer, oral solution..
  Arms: Part B (multiple ascending dose) ADME
Drug: Microtracer matching placebo (MAD - ADME) — Single dose of 14C-ACT-777991 microtracer matching placebo, oral solution.
  Arms: Part B (multiple ascending dose) ADME

SUMMARY:
A study to examine the safety, tolerability, and pharmacokinetics of single- and multiple-ascending doses of ACT-777991 in healthy subjects.

ELIGIBILITY:
General Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male (Part A and B) and female subjects (Part B) aged between 18 and 55 years (inclusive) at Screening.
* Healthy on the basis of medical history, physical examination, cardiovascular assessments, and clinical laboratory tests.
* Male subjects with a partner who might become pregnant must either be vasectomized or agree to practice adequate contraception from admission to the study site until 3 months after dosing, or the partner must consistently and correctly use a highly effective method of contraception.

Inclusion Criteria for Part B:

* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use a highly effective method of contraception with a failure rate of less than 1% per year, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.

General Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment.

Exclusion Criteria for the absorption,distribution, metabolism and excretion (ADME) evaluation:

* Radiation exposure, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 milli sievert (mSv) in the last 12 months or 10 mSv in the last 5 years. Occupationally exposed workers, as defined in the relevant Ionising Radiation Regulations, must not participate in the study.
* Participation in any study involving administration of any Carbon-14 (14C) radiolabeled compound within the 12 months prior to Screening.

Exclusion Criteria for Part B:

* Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events. | From first dose on Day 1 to Day 4 after the last dose was administered

SECONDARY OUTCOMES:
All cohorts: Area under the plasma concentration-time curve (AUC) from zero to time t of the last measured concentration above the limit of quantification (AUC0-t) of ACT-777991 | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
All cohorts: Area under the plasma concentration-time curve (AUC) from zero to infinity (AUC0-inf) of ACT-777991 | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
All cohorts: Maximum plasma concentration (Cmax) of ACT-777991 | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
All cohorts: Time to reach Cmax (tmax) of ACT-777991 | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
All cohorts: Terminal half-life (t1/2) of ACT-777991 | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
Part A (SAD): Absolute bioavailability of ACT-777991 | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
Part B (MAD): Excretion of radioactivity in urine and feces | Samples will be collected at predefined time points from Day 1 to Day X+3 (where Day X = day of last study treatment administration)
Part B (MAD): AUC during a dosing interval (AUCτ) following the first and the last dose of ACT-777991. | Blood samples will be collected at predefined time points from Day 1 to Day 4 after the last dose was administered
Part A (SAD): Food effect evaluation only: AUC0-inf of ACT-777991 under fed conditions | Blood samples will be collected at predefined time points from Day 1 to Day 4.
Part A (SAD): Food effect evaluation only: Cmax of ACT-777991 under fed conditions | Blood samples will be collected at predefined time points from Day 1 to Day 4.
Part A (SAD): Food effect evaluation only: tmax of ACT-777991 under fed conditions | Blood samples will be collected at predefined time points from Day 1 to Day 4.
Part A (SAD): Food effect evaluation only: t1/2 of ACT 777991 under fed conditions | Blood samples will be collected at predefined time points from Day 1 to Day 4.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No